CLINICAL TRIAL: NCT01758445
Title: Phase II Study of Postoperative, Cardiac-Sparing Proton Radiotherapy for Patients With Stage II/III,Loco-Regional, Non-Metastatic Breast Cancer Requiring Whole Breast or Chest Wall Irradiation With Lymph Node Irradiation
Brief Title: Proton Radiation for Stage II/III Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Proton Collaborative Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRE008-12
Record Dates: First submitted 2012-12-14; First posted 2013-01-01 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast Neoplasm; Breast Tumor; Cancer of the Breast
Keywords: Breast; Cancer; Radiation; Proton
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Radiotherapy (Experimental): Proton Radiotherapy
  Interventions: Radiation: Proton Radiotherapy

INTERVENTIONS:
Radiation: Proton Radiotherapy — Radiation therapy will be given once a day. Minimum of 28 treatments and may receive 6-9 additional treatments as determined by protocol & physician.

SUMMARY:
The purpose of this study is to look at the rates of acute and long term adverse events of postoperative proton radiotherapy for complex loco-regional irradiation in women with loco-regionally advanced breast cancer. This study specifically includes longitudinal follow up to assess the incidence of cardiac mortality and second malignant neoplasms at 10 and 15 years following proton therapy(PT).

DETAILED DESCRIPTION:
The proposed Phase II study is seeking to build clinical data as a continuation of the original dosimetric analysis published by Ares et al. performed at Paul-Scherrer Institute (PSI). That comparison demonstrated a benefit form proton planning for patients with non-metastatic breast cancer requiring complex, loco-regional, postoperative radiotherapy.1 The advantages of PT were improved target coverage compared to standard photon irradiation and reduced dose to heart, lungs and contralateral breast.

The study goal is to demonstrate a "meaningful benefit" of proton therapy for women with loco-regionally advanced breast cancer. The main clinical endpoints of this trial are the reduction of cardiac morbidity and mortality (coronary artery disease, myocardial infarction, cardiac insufficiency) and the reduction of contralateral, second breast cancer. Both adverse events are presently associated with external beam photon therapy. Both goals require longitudinal follow-up of minimum 5-10 years. Despite the logistical challenges of long term follow-up, the effort is needed in view of the compelling preclinical evidence of dose avoidance or even absence of radiation dose to heart and contralateral breast uniquely accomplishable by protons only.

ELIGIBILITY:
Inclusion Criteria:

1. Must sign study-specific, IRB approved informed consent form prior to study entry. Note consent by legally authorized representative is not allowed for this trial.
2. Must be > = 18 years of age.
3. Must have a life expectancy of at least 10 years based on age and comorbidities but excluding diagnosis of breast cancer.
4. Must have pathology proven breast cancer. Pathology must be invasive ductal or lobular
5. Must meet stage II - III group criteria per AJCC Staging manual 7th edition.
6. Must have had surgical treatment of the breast - either mastectomy or breast preserving surgery, such as lumpectomy. Re-excision of surgical margins is permitted.
7. Note: Multicentric breast cancer and Paget's disease of the nipple are permitted.

Exclusion Criteria:

1. Weight over 410 pounds.
2. Non-epithelial breast malignancies such as sarcoma or lymphoma.
3. Surgical margins that cannot be microscopically assessed or are positive at pathologic evaluation. (If surgical margins are rendered free of disease by re-excision, the patient is eligible).
4. Breast size exceeding the technical limitation of daily set-up reproducibility. This may be center-specific and will be assessed at the discretion of the treating center.
5. Women with post-surgical temporary breast expanders will require individual assessment. Depending on the manufacturing product and other treatment planning-specific details the patient may be eligible or may be deemed ineligible, as determined by treating investigator.
6. Prior history of breast cancer.
7. Prior radiation to the breast or thorax.
8. Collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma.
9. Pregnancy or lactation at the time of proposed study entry. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy such as an intrauterine device or condom with spermicide. (Note: Women of childbearing potential must have a negative serum pregnancy test within 3 weeks of study registration).
10. Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
11. Prior history of non-breast malignancies unless they have been disease free for 5 or more years and are deemed by their physician to be at low risk for recurrence. Further, patients who have the following cancers treated within the prior 5 years are permitted: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-02; Primary Completion 2027-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the rates of acute and late toxicities (acute and late adverse events) resulting from proton therapy radiation treatment. | 5 years

SECONDARY OUTCOMES:
Compare dosimetrically the dose volume histogram (DVH) of the PT plans with conventional external beam plans (either photon/electron intensity modulated radiotherapy(IMRT)plans, 3D-photon plans, or Tomotherapy plans). | On average at 9 weeks post start of treatment
Incidence rates of local control, regional control, metastatic status and disease free overall survival. | 5 years
Compare the different DVH parameters for the targets (D2, Dmean, Dmin, D95, V95, V110) and different OARs (as described later) of the PT plans with the corresponding values of the 3D-conformal radiation therapy (CRT), IMRT and Tomotherapy plans. | On average at 9 weeks post start of treatment
Determine dose distribution of proton therapy to coronary arteries, heart, ipsilateral and contralateral lung, and contralateral breast. | On average at 9 weeks post start of treatment
Determine the incidence of clinically symptomatic coronary artery disease, cardiac morbidity and mortality in general and incidence of secondary malignancy, including contralateral breast cancer | 5 years
Evaluate quality of life results. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eugen Hug, MD, Study Chair — Proton Collaborative Group
Locations (5):
- United States (5):
  - Northwestern Medicine Chicago Proton Center, Warrenville, Illinois
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - Princeton ProCure Managment LLC, Somerset, New Jersey
  - Oklahoma Proton Center, Oklahoma City, Oklahoma
  - Hampton University Proton Therapy Institute, Hampton, Virginia